CLINICAL TRIAL: NCT01041326
Title: A Phase I Dose-Escalation Study of Preoperative Radiation Therapy Followed by Radical Prostatectomy in Patients With High Risk, Localized Carcinoma of the Prostate
Brief Title: Preoperative Radiation Therapy for High Risk Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006510
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; radiation; neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Leve 1 Radiation (Experimental): Subjects in Group 1 will receive 39.6 Gy (at 1.8 Gy/fx) to the whole pelvis. The subject will then undergo radical prostatectomy between 4-8 weeks after completion of radiation.
  Interventions: Radiation: Radiation; Procedure: Radical Prostatectomy
- Level 2 Radiation (Experimental): Subjects in Group 2 will receive 45 Gy (at 1.8 Gy/fx) to the whole pelvis. The subject will then undergo radical prostatectomy between 4-8 weeks after completion of radiation.
  Interventions: Radiation: Radiation; Procedure: Radical Prostatectomy
- Level 3 Radiation (Experimental): Subjects in Group 3 will receive 45 Gy to the whole pelvis, followed by a boost to the prostate and periprostatic tissue, for total doses of 50.4 Gy. The subject will then undergo radical prostatectomy between 4-8 weeks after completion of radiation.
  Interventions: Radiation: Radiation; Procedure: Radical Prostatectomy
- Level 4 Radiation (Experimental): Subjects in Group 4 will receive 45 Gy to the whole pelvis, followed by a boost to the prostate and periprostatic tissue, for total doses of 54 Gy. The subject will then undergo radical prostatectomy between 4-8 weeks after completion of radiation.
  Interventions: Radiation: Radiation; Procedure: Radical Prostatectomy

INTERVENTIONS:
Radiation: Radiation — Pre-operative Radiation to Prostate, SV, and Pelvic Lymph Nodes
Procedure: Radical Prostatectomy — Patients will undergo evaluation by a surgeon for consideration of resection after completion of radiation therapy. If a surgical resection is possible, it is recommended that patients undergo surgery four to eight weeks after completion of radiation therapy. This surgical procedure will be performed by one of the standard accepted approaches.

SUMMARY:
This is a Phase I dose-escalation study of moderate dose radiation therapy prior to radical prostatectomy for patients with high-risk localized disease. Its hypothesis is that such treatment will be well tolerated with similar side effect profile as surgery alone. Patients in Groups 1 and 2 will receive 39.6 Gy and 45 Gy (at 1.8 Gy/fx), respectively, to the whole pelvis. Patients in Groups 3 and 4 will receive 45 Gy to the whole pelvis, followed by a boost to the prostate and periprostatic tissue, for total doses of 50.4 and 54 Gy, respectively. The patient will then undergo radical prostatectomy between 4-8 weeks after completion of radiation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have

* biopsy-confirmed "high-risk" prostate cancer, defined as A. PSA > 20, B. Gleason Score (GS) >/= 8, and/or C. Clinical stage T3 disease per AJCC Staging Manual, 6th edition; or D. At least two out of three of the following: PSA 10-19.9, GS = 7, or clinical stage = T2b / T2c.
* a negative bone scan,
* be medically fit to undergo surgery as determined by treating urologist,
* age > 18,
* KPS must be >/= 80,
* no prior pelvic radiation therapy, chemotherapy, or androgen deprivation,
* no prior invasive malignancy, except non- melanomatous skin cancer unless disease free for a minimum of 5 years. Carcinoma in-situ of the bladder or head and neck region is permissible.
* Subjects must freely sign informed consent to enroll in the study.

Exclusion Criteria:

* prior pelvic radiation therapy, chemotherapy, or androgen deprivation,
* prior invasive malignancy, except non- melanomatous skin cancer, carcinoma in-situ of the bladder or head and neck region, unless disease free for a minimum of 5 years.
* Metastatic disease as demonstrated by bone scan, CT scan or MRI of the pelvis, or chest x-ray.
* Pathologically documented positive pelvic lymph nodes. If Pre-operative CT scan or MRI (ordered at the discretion of the treating physicians) demonstrates lymph nodes which are suspicious for involvement, then biopsy must be undertaken and nodes proven negative before patient can enroll on this trial.
* Declared high-risk for anesthesia by attending anesthesiologist, cardiologist, or other physician.
* History of prior pelvic radiation therapy.
* History of androgen deprivation therapy or chemotherapy.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
post-operative morbidity | 30 day

SECONDARY OUTCOMES:
continence | 1 year
erectile function | 1 year
biochemical recurrence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bridget F Koontz, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Koontz BF, Quaranta BP, Pura JA, Lee WR, Vujaskovic Z, Gerber L, Haake M, Anscher MS, Robertson CN, Polascik TJ, Moul JW. Phase 1 trial of neoadjuvant radiation therapy before prostatectomy for high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2013 Sep 1;87(1):88-93. doi: 10.1016/j.ijrobp.2013.05.014. Epub 2013 Jun 19. PMID 23790772